CLINICAL TRIAL: NCT02106260
Title: A Phase I/IIa Open-label First-in-Human Study to Assess Safety and Pharmacokinetics and Explore Biomarker Effects of Topical Ionic Contra-viral Therapy (ICVT) Comprised of CLS003 in Subjects With Cutaneous Warts
Brief Title: First-in-Human Study of CLS003 ICVT in Subjects With Cutaneous Warts
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLS003-CO-PR-001
Record Dates: First submitted 2014-04-02; First posted 2014-04-08 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Cutaneous Warts
Keywords: safety; pharmacokinetics (PK); pharmacodynamics (PD); CLS003

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CLS003 (Experimental)
  Interventions: Drug: CLS003

INTERVENTIONS:
Drug: CLS003

SUMMARY:
This phase I/IIa study has an open-label, First-in-Human (FIH), single center design to assess the safety, pharmacokinetics (PK) and pharmacodynamics (PD) of multiple doses of topically applied CLS003 in healthy subjects with cutaneous warts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (male, non-pregnant female), 18 to 65 years of age, inclusive.
* Body mass index (BMI) between 18 and 30kg/m2, inclusive
* Fitzpatrick skin type I-II-III-IV
* At least 4 cutaneous warts on the hands, separated by at least 1cm of skin

Exclusion Criteria:

* For women, a positive pregnancy test and/or nursing at screening
* A positive test for drugs of abuse at screening
* History of alcohol or illicit drug abuse
* Positive test results for Hepatitis B, Hepatitis C or HIV
* Have used salicylic acid or any other over-the-counter- wart-removing product in the treatment area within 30 days prior to enrollment
* Have received cryotherapy in the treatment area within 60 days prior to enrollment
* Have required systemic intake of immunosuppressive or immunomodulatory medication (including oral or parenteral corticosteroids) with 30 days prior to enrollment or during the course of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of CLS003 | 7 days
Number of participants with adverse events | 7 days
Peak Plasma Concentration (Cmax) of CLS003 | 7 days
Time to reach Cmax (Tmax) | 7 days

SECONDARY OUTCOMES:
Pharmacodynamic effects of topically applied CLS003 on wart morphology and HPV viral load | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: J. (Koos) Burggraaf, MD, PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Zernikedreef 8, Netherlands